CLINICAL TRIAL: NCT03622866
Title: Clinical Trial Comparing Ultra-High Versus Traditional Pulse Widths Using the ALGOVITA® SCS System High Fidelity Stimulation in the Treatment of Persistent or Recurrent Back and/or Leg Pain Following Spinal Surgery
Brief Title: Algovita Spinal Cord Stimulation System Hi-Fi Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor bankruptcy
Sponsor: Nuvectra (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CLRE 1092
Record Dates: First submitted 2018-07-26; First posted 2018-08-09 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: During the Treatment Phase of the study, all subjects will receive both treatments under a crossover design. Subjects will undergo 12 weeks of treatment in each group with a 1-week washout between groups.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects who receive a permanent implant will be randomly assigned in a 1:1 ratio to one of the two sequences of treatment. Randomization schedules for each site will be prepared by the contract research organization (CRO) statistician and uploaded into a role-limited module of the study database. In order to avoid any potential bias, each site will designate an unblinded coordinator (UC). The UC, Nuvectra field personnel (FP) and the CRO will be unblinded to the treatment group. The participant and other site staff will be blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ultra-high pulse width (Active Comparator): Ultra-high pulse width stimulation using the Algovita System
  Interventions: Device: Ultra-high pulse width stimulation
- Traditional pulse width (Active Comparator): Traditional pulse width stimulation using the Algovita System
  Interventions: Device: Traditional pulse width stimulation

INTERVENTIONS:
Device: Ultra-high pulse width stimulation — Algovita Spinal Cord Stimulation System with associated components
  Arms: Ultra-high pulse width
Device: Traditional pulse width stimulation — Algovita Spinal Cord Stimulation System with associated components
  Arms: Traditional pulse width

SUMMARY:
The objective of this study is to obtain post-market clinical outcome data for the Algovita SCS System when used on-label, according to the applicable directions for use, using high fidelity tonic stimulation at either ultra-high pulse width or traditional pulse width for the treatment of persistent or recurrent back and/or leg pain following spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FBSS defined as persistent or recurrent back and/or leg pain despite one or more anatomically successful back surgeries for the same original pain.
* Age 18-75 years old at consent.
* Targeted pain intensity of ≥ 5 out of 10 on the Baseline visit NRS.
* ODI score of 41-80 out of 100 at the Baseline visit.
* Appropriate candidate for the surgical procedure and Algovita SCS therapy based on the clinical judgment of the investigator and the Algovita Instructions for Provider (IFP) in the Nuvectra product manuals.
* On stable pain medications for at least 28 days prior to consent. Stable is defined as no new or discontinued pain medications and no changes to total daily dose of any pain medications.
* Willing and capable of providing informed consent.
* Willing and able of complying with the study-related requirements, procedures, and visits.
* Speaks English as a primary language (as the Algovita patient manuals are only currently available in English).
* Has adequate cognitive ability to use the subject devices (e.g., PPC, PoP), as determined by the investigator.

Exclusion Criteria:

* Has a medical/psychological/psychiatric condition/disorder that could interfere with study procedures as determined by the investigator.
* Has a coexisting pain condition that might confound pain ratings, as determined by the investigator.
* Has a condition currently requiring or likely to require the use of MRI or diathermy.
* Has an existing drug pump, SCS System, or other active implantable device.
* Has any prior SCS experience.
* Pregnant or planning to become (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile, or be at least 2 years postmenopausal).
* For subjects with diabetes, HbA1c ≥ 8.5% as measured at the Baseline visit (or within the 3 months prior to the Baseline visit).
* Participating in another clinical trial that could affect the outcomes or requirements of this study as determined by the investigator.
* Involved in an injury claim under current litigation or have a pending or approved workers compensation claim.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Effectiveness of targeted pain reduction compared to baseline in each treatment arm | Week 25
  The percentage of participants who experience at least a 50 percent reduction in targeted pain from baseline, as assessed by Numeric Rating Scale (NRS). The Numeric Rating Scale (NRS) will range from 0 to 10 with a higher score indicating a higher level of pain.
  Effectiveness will be compared both descriptively and statistically between the two randomized treatment groups using crossover analysis methods.
Rate of serious study-related adverse events (AEs) in each treatment arm | From Permanent Implant through Week 25
  The rate of serious study-related AEs. Study-related AEs are defined as any device, procedure and therapy/stimulation-related AEs.

SECONDARY OUTCOMES:
Effectiveness of targeted pain reduction compared to baseline in each treatment arm | Week 12 and Months 12, 18 and 24
  The percentage of participants who experience at least a 50 percent reduction in targeted pain as assessed by Numeric Rating Scale (NRS). The Numeric Rating Scale (NRS) will range from 0 to 10 with a higher score indicating a higher level of pain.
Effectiveness of back and/or leg pain reduction compared to baseline in each treatment arm | Weeks 12 and 25, and Months 12, 18 and 24
  The percentage of participants who experience at least a 50 percent reduction in back and/or leg pain as assessed by Numeric Rating Scale (NRS). The Numeric Rating Scale (NRS) will range from 0 to 10 with a higher score indicating a higher level of pain.
Effectiveness of targeted, back and/or leg pain reduction compared to baseline in each treatment arm | Weeks 12 and 25, and Months 12, 18 and 24
  The percentage of participants who experience at least a 50 percent reduction in targeted, back and/or leg pain as assessed by a Visual Analog Scale (VAS). The Visual Analog Scale (VAS) will range from 0 mm (no pain) to 100 mm (worst pain imaginable). A higher score indicates a higher level of pain.
Change in targeted, back and/or leg pain compared to baseline in each treatment arm | Weeks 12 and 25, and Months 12, 18 and 24
  The mean change and percent change from baseline in targeted, back and/or leg pain as assessed by a Numeric Rating Scale (NRS). The Numeric Rating Scale (NRS) will range from 0 to 10 with a higher score indicating a higher level of pain.
Change in targeted, back and/or leg pain compared to baseline in each treatment arm | Weeks 12 and 25, and Months 12, 18 and 24
  The mean change and percent change from baseline in targeted, back and/or leg pain as assessed by a Visual Analog Scale (VAS). The Visual Analog Scale (VAS) will range from 0 mm (no pain) to 100 mm (worst pain imaginable). A higher score indicates a higher level of pain.
Clinician Global Impression of Change score in each treatment arm | Weeks 12 and 25, and Months 12, 18 and 24
  The Investigator's assessment of change in the overall status of the participant using the standard Clinician Global Impression of Change ranging from 1 (very much improved) to 7 (very much worse).
Change in disability compared to baseline in each treatment arm | Weeks 12 and 25, and Months 12, 18 and 24
  The change from baseline in disability as measured by the Oswestry Disability Index. The Oswestry Disability Index is scored between 0 and 100 with higher scores indicating a greater disability.
Change in quality of life compared to baseline in each treatment arm | Weeks 12 and 25, and Months 12, 18 and 24
  The change from baseline in quality of life as measured by the EQ-5D-5L, a standardized measure of health status.
Change in patient activity per the Pain Disability Index score in each treatment arm | Weeks 12 and 25, and Months 12, 18 and 24
  The change from baseline in patient activity as measured by the Pain Disability Index score. The Pain Disability Index is a self-report asking participants to rate how much pain interferes in seven areas of life activity using a 0 (no disability) to 10 (total disability) numeric rating scale.
Patient Global Impression of Change score in each treatment arm | Weeks 12 and 25, and Months 12, 18 and 24
  The participant's assessment of change in their overall status using the standard Patient Global Impression of Change ranging from 1 (very much improved) to 7 (very much worse).
Participant satisfaction per the subject satisfaction survey outcome in each treatment arm | Weeks 12 and 25, and Months 12, 18 and 24
  Participant satisfaction using a subject satisfaction survey (5 point Likert scale format) ranging from very satisfied to very dissatisfied.
Evaluation of trial success rates | From Trial Implant to End of Trail
  The percentage of participants that have a successful trial phase, defined as at least a 50 percent reduction in targeted pain compared to baseline.
Rate of surgical re-intervention of the SCS system | From Permanent Implant through Month 24
  Rate of surgical re-intervention of the SCS system for participants with a permanent implant.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Tranchina, Study Director — Nuvectra
Locations (10):
- United States (10):
  - Pain Institute of Southern Arizona, Tucson, Arizona
  - Newport Beach Headache & Pain, Newport Beach, California
  - Summit Pain Alliance, Santa Rosa, California
  - Spinal Diagnostics & Pain Management, Colorado Springs, Colorado
  - Mid-America PolyClinic & Interventional Pain Management Specialists, Overland Park, Kansas
  - WK River Cities Clinical Research Center, Shreveport, Louisiana
  - Brigham & Women's Hospital, Chestnut Hill, Massachusetts
  - Adena Spine Center, Chillicothe, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Comprehensive Spine Center at Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No